CLINICAL TRIAL: NCT01655030
Title: A Double-Blind, Randomized, Placebo-Controlled Clinical Trial to Evaluate the Efficacy of Creatine Monohydrate as Adjunctive Therapy for Bipolar Depression
Brief Title: Creatine Monohydrate as Adjuvant Therapy for Bipolar Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alexandre Toniolo, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR-BD-RCT
Record Dates: First submitted 2012-07-29; First posted 2012-08-01 (Estimated); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Bipolar I Disorder; Current Episode Depressed
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- creatine monohydrate (Experimental): 6g qd for 6 weeks
  Interventions: Dietary Supplement: creatine monohydrate
- placebo (Placebo Comparator): 6g qd for 6 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: creatine monohydrate
  Arms: creatine monohydrate
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether creatine monohydrate is effective as an adjuvant treatment for bipolar depression.

DETAILED DESCRIPTION:
Bipolar Depression is associated with high rates of disability and increased mortality. Despite its major negative impact, treatment of Bipolar Depression is still controversial and only partially efficacious, with over half of patients not responding adequately to available treatment. In this context, the use of drugs that modulate energy metabolism has been proposed as promising new option as treatment strategies for bipolar depression. The aim of our proposed study is to perform a 6-week randomized, double-blind, placebo-controlled clinical trial of creatine monohydrate as an adjuvant treatment for bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Individuals eligible for the study will be adults aged 18 to 60 years of age who met DSM-IV criteria assessed by the SCID (Structural Clinical Interview for DSM-IV) for type I bipolar disorder, current episode depressed.
* Patients who have scored > 19 on the Montgomery-Asberg Depression Rating Scale (MADRS) will be included, although more than two weeks of treatment with lithium (serum level> 0.8 mEq / L), valproate (serum levels> 50 mg / L) or quetiapine (300-600mg/dia dose) or drug combination.
* Antipsychotics, anticonvulsants, benzodiazepines, and thyroid supplementation will be allowed if the dose has remained stable over the past two weeks.
* Antidepressants will be allowed if the dosage has remained stable for 4 weeks.

Exclusion Criteria:

* Subjects with substance abuse within 2 weeks before inclusion or substance dependence up to 2 months will not be included.
* Other exclusion criteria will be:

  * diagnosis of schizophrenia,
  * dementia,
  * delirium,
  * epilepsy,
  * mental retardation,
  * clinically unstable medical illnesses,
  * preexisting renal disease,
  * history of hypersensibility to creatine.
* Not included are individuals at high risk for suicidal or homicidal behavior or self-mutilation will not be included.
* Women with gestational potential can only be included if they are using reliable contraception.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
MADRS (Montgomery-Asberg Depression Rating Scale) | 6 weeks
  change of score on the Montgomery-Asberg Depression Rating Scale

SECONDARY OUTCOMES:
HDRS-17 (Hamilton Depression Rating Scale - 17-item version) | 6 weeks
  change of score on the Hamilton Depression Rating Scale - 17-item version

OTHER OUTCOMES:
CGI (Clinical Global Impressions Scale) - Severity and Improvement | 6 weeks
  change of score on the Clinical Global Impressions Scale
YMRS (Young Mania Rating Scale) | 6 weeks
  change of score on the Young Mania Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Beny Lafer, PhD, Principal Investigator — Bipolar Disorder Research Program, Coordinator, IPq-HC-FMUSP
Locations (1):
- Institute of Psychiatry - HC-FMUSP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Toniolo RA, Silva M, Fernandes FBF, Amaral JAMS, Dias RDS, Lafer B. A randomized, double-blind, placebo-controlled, proof-of-concept trial of creatine monohydrate as adjunctive treatment for bipolar depression. J Neural Transm (Vienna). 2018 Feb;125(2):247-257. doi: 10.1007/s00702-017-1817-5. Epub 2017 Nov 24. PMID 29177955